CLINICAL TRIAL: NCT03494231
Title: An Open-label, Dose Escalation Phase 1 Study to Investigate HLX06, a Humanized Monoclonal Antibody Targeting Human Vascular Endothelial Growth Factor Receptor-2, in Patients With Advanced Solid Tumors Refractory to Standard Therapy
Brief Title: A Study of HLX06, a Humanized Monoclonal Antibody Targeting Human Vascular Endothelial Growth Factor Receptor-2 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Henlix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX06-001
Record Dates: First submitted 2018-03-11; First posted 2018-04-11 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumor, Adult
Keywords: Metastatic; Refractory; Cancer; Solid; Tumor
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Intervention Model Description: The modified accelerated titration design (ATD) 2A and Bayesian optimal interval design (BOIN)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HLX06, in patients with solid cancers (Experimental): Each cycle of treatment consists of 4 weeks. Patients who enroll into this study will receive an infusion of assigned dose of HLX06 once per week. No intra-patient dose escalation is allowed. The proposed dose escalation sequence is 500, 750, 900, 1200, 1500 mg, starting from 500 mg/kg.
  Interventions: Drug: HLX06

INTERVENTIONS:
Drug: HLX06 — recombinant fully human anti-VEGFR2 monoclonal antibody against cancers
  Other Names: anti-VEGFR2 monoclonal antibody

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of fully human anti-VEGFR2 monoclonal antibody, HLX06, in patients with advanced or metastatic tumors refractory to standard therapy. This study will also evaluate the pharmacokinetics, pharmacodynamics, immunogenicity and anti-tumor effect of HLX06 and explore the potential prognostic and predictive biomarkers.

DETAILED DESCRIPTION:
Angiogenesis plays an important role in cancer development. The VEGF family and their receptors (VEGFR) are well characterized for their role in neoplastic angiogenesis. VEGFR2 belongs to type V receptor tyrosine kinase encoded by KDR gene, and is expressed in vascular endothelial cells. It is a primary responder to vascular endothelial growth factor signal that regulates endothelial migration and proliferation. The expression of VEGFR2 can be found in multiple tumor types, including angiosarcoma, Kaposi sarcoma. In epithelial carcinoma, VEGFR2 expression can be found in mesothelioma, non-small cell lung cancer, and embryonal carcinoma. Targeting angiogenesis using either small molecule inhibitors or biological agents have been widely used in current cancer management. Current approved anti-angiogenesis biological agents include bevacizumab, ramucirumab, aflibercept. Among them, ramucirumab (IMC-1121B) targets vascular endothelial growth factor receptor 2 (VEGFR2). Ramucirumab has been approved for use in combination with paclitaxel for second-line treatment of patients with advanced gastric or gastroesophageal junction adenocarcinoma.

Although ramucirumab has been approved for gastric cancer, its improvement in overall survival is still not satisfactory. It prolongs the overall survival by 6 weeks when combined with paclitaxel. So far, there is not biomarker available to predict the efficacy of ramucirumab. Therefore, a new monoclonal antibody also targeting VEGFR2 might provide better efficacy for cancer patients.

HLX06 is a new, fully human monoclonal antibody targeting VEGFR2. It has better binding affinity to VEGFR2, and also binds to different region in VEGFR2. In vitro studies have demonstrated the growth inhibition of human endothelial cells, and HLX06 has shown growth inhibition of tumors in xenogeneic studies.

Nonclinical studies up to weekly 150 mg/kg in cynomolgus monkeys for 13 weeks have shown good tolerability without evident toxicities (please refer to Investigator's brochure). HLX06 shows cross-reactivity to both monkey and human VEGFR2, but does not bind rodent VEGFR2. The investigators expect that HLX06 will provide a better alternative than ramucirumab for patients with advanced cancers.

However, HLX06 has not yet been tested in humans. Therefore, the investigators propose this first-in-human phase 1 study. In this study, the investigators intend to monitor the safety and tolerability of HLX06 in humans, and hope to identify the maximum tolerated dose, and determine the recommended phase 2 dose for future study. At the same time, the investigators would like to collect information of the pharmacokinetics and pharmacodynamics of this drug and its potential immunogenicity.

To minimize the risk of patients who volunteer to receive this experimental drug, the investigators have selected 250 mg flat dose as the starting dose. The reason for using flat dosing instead of body weight-adjusted dosing is based on previous population pharmacokinetic studies for multiple monoclonal antibody drugs. The 500 mg flat dose was conservatively selected to provide sufficient safety factor in the FIH study, based on 1/6 of the human equivalent dose (1/3) of the highest non-severely toxic dose (HNSTD) in 3 month repeat-dose studies in cynomolgus monkeys.

To investigate the dose required to reach maximal effect, the investigators propose a dose escalation sequence. The purpose of the dose escalation is to obtain the pharmacokinetics and pharmacodynamics of HLX06 at different dose levels, and investigate its relationship with adverse reactions. Also, the investigators intend to identify the MTD. The information from the dose escalation is crucial to determine the optimal dose in future studies and potential indications for HLX06.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed, unidimensionally-measurable and/or evaluable carcinoma which has failed standard therapy or for whom no standard therapy is available.
2. ECOG performance status score of ≤ 2 at study entry.
3. Able to provide written informed consent.
4. Adequate hematologic functions, as defined by: absolute neutrophil counts ≥ 1500/mm3; a hemoglobin level ≥ 10 gm/dL; a platelet count ≥ 100,000/mm3.
5. Adequate hepatic function defined by: a total bilirubin level ≤ 1.5x of upper limit of normal (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2.5x of ULN or ≤ 5x of ULN in known hepatic metastases or with primary hepatocellular carcinoma.
6. Adequate renal function, as defined by the creatinine clearance rate ≥ 50 mL/minute by Cockcroft-Gault formula.
7. Adequate cardiac function defined as left ventricular ejection fraction (LVEF)≥ 50%.
8. Use of effective contraceptive measures if procreative potential exists.
9. At least 28 days from prior major surgery, prior cytotoxic chemotherapy, or prior therapy with investigational agents (or medical device) or local radiotherapy before 1st infusion of HLX06.
10. For patients with hepatocellular carcinoma, their Child-Pugh score has to be A.
11. Able to be followed up as required by the study protocol.

Exclusion Criteria:

1. Patients with large centrally located pulmonary lesions adjacent to or invading large blood vessels.
2. Hemoptysis more than ½ teaspoon (approximately 2-3 mL) of red blood per day.
3. Patients who still have ≥ grade 2 toxicities from prior therapies.
4. Concurrent unstable or uncontrolled medical conditions with either of the followings:

   * Active systemic infections;
   * Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg), or poor compliance with anti-hypertensive agents;
   * Clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (class III or IV of New York Heart Association [NYHA]) or acute myocardial infarction within 6 months;
   * Uncontrolled diabetes or poor compliance with hypoglycemics;
   * The presence of chronically unhealed wound or ulcers
   * Other chronic diseases, which, in the opinion of the investigator, could compromise safety of the patient or the integrity of study.
5. Newly-diagnosed or symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not taking steroids for brain edema). Anticonvulsants are allowed.
6. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 3 years are allowed to participate).
7. Pregnancy (confirmed by serum beta human chorionic gonadotropin [ßHCG]) or breast-feeding (for female patients only).
8. A known history or clinical evidence of a deep vein or arterial thrombosis, or pulmonary embolism within 6 months of first infusion of HLX06.
9. Less than six weeks from last infusion of ramucirumab, or any other anti-VEGF monoclonal antibody therapy (Last treatment with other monoclonal antibodies targeting proteins other than anti-angiogenic factors is permitted if ≥ 4 weeks prior to the first infusion of HLX06).
10. Proteinuria ≥ 2+ in routine urinalysis (patients with a protein value of ≤500 mg confirmed by a 24-hour urine collection are eligible).
11. Known history of human immunodeficiency virus infection (HIV).
12. The patient is the investigator, sub-investigator or any one directly involved in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tus-Yi Chao, MD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03494231/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03494231/ICF_001.pdf